CLINICAL TRIAL: NCT03721679
Title: Poly-ICLC (Hiltonol®) Plus Anti-PD1 or Anti-PD-L1 in Unresectable Solid Cancers An Adaptive Phase I/II Clinical Pilot Study
Brief Title: Poly-ICLC (Hiltonol) and Anti-PD1 or Anti-PD-L1
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Recruiting target patients is intermittent making it impracticable to enroll the required study sample. The administrative responsibilities have been met with extraordinary challenges. Current funding does not match the incurring costs.
Sponsor: Oncovir, Inc. (Industry)
Collaborators: Chevy Chase Healthcare, Chevy Chase MD (Unknown); Mt. Sinai School of Medicine, New York, New York (Unknown); Bay Hematology Oncology PA, Easton MD (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ONC2018-001
Record Dates: First submitted 2018-10-01; First posted 2018-10-26 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2020-12

CONDITIONS: Solid Cancer
Keywords: Immunotherapy; Vaccine Therapy
MeSH Terms: interventions — Nivolumab; pembrolizumab; atezolizumab; durvalumab; S-Adenosylmethionine

STUDY DESIGN:
Intervention Model Description: The study is largely a signal-finding exercise to determine if there is an immune and/or clinical response to the addition of poly-ICLC to aPD-1 or aPDL-1 therapy, as predicted by preclinical models.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Poly-ICLC treatment combination aPD-1or aPD-1L1 (Experimental): Weeks 1 and 2: Poly-ICLC (Hiltonol®) 1 mg (0.5 ml) IM ONLY twice a week with a 48-72 hour interval between the two injections
  Weeks 3-25:
  1. Poly-ICLC (Hiltonol®) 1 mg (0.5 ml) IM twice a week with a 48-72 hour interval between the two injections, AND
  2. ONLY 1 of the following regimens will be administered, per manufacturer's dosing and clinical oncologist's discretion as follows:
     * Nivolumab (Opdivo), OR
     * Pembrolizumab (Keytruda), OR
     * Cemiplimab (Libtayo) OR
     * Atezolizumab (Tecentriq) OR
     * Durvalumab (Imfinzi) Follow up: After completion of treatment subjects may be contacted by telephone at least twice over 12 months, or longer with patient consent, in order to inquire on their health status (e.g., in remission, progressive disease, on new cancer treatment).
  Interventions: Biological: Poly-ICLC combination treatment with aPD-1 (Nivolumab or Pembrolizumab) or aPD-L1 (Atezolizumab or Durvalumab) over 6 months

INTERVENTIONS:
Biological: Poly-ICLC combination treatment with aPD-1 (Nivolumab or Pembrolizumab) or aPD-L1 (Atezolizumab or Durvalumab) over 6 months — Same as above
  Other Names: Same as above

SUMMARY:
This is an open labeled, non-randomized adaptive pilot study. The study interventions involved in this study are:

Poly-ICLC (Polyinosinic-Polycytidylic acid stabilized with polylysine and carboxymethylcellulose, also known as Hiltonol®) treatment in combination with anti-PD-1 (Nivolumab, Cemiplimab or Pembrolizumab) or anti-PD-L1 (Atezolizumab or Durvalumab)

DETAILED DESCRIPTION:
This research study is a PhaseI/II clinical trial investing a combination of targeted therapies as possible treatment for advanced solid cancers

FDA has not yet approved Poly-ICLC as treatment for diseases in this study

Pembrolizumab, Nivolumab, Atezolizumab, Cemiplimab and Durvalumab are now FDA approved for certain patients with multiple cancer types.

The study is designed to evaluate the safety of intramuscular (IM) Polyinosinic-polycytidylic acid stabilized with polylysine and carboxymethylcellulose (Poly-ICLC, Hiltonol®) in combination with Anti-PD-1 or Anti-PD-L1 for treatment of study subjects with advanced solid cancers.

ELIGIBILITY:
Inclusion Criteria

1. Histologically confirmed diagnosis of Solid Cancer, independent of PD-L1 tumor status.
2. Patients must be 18 years of age or older.
3. Unresectable disease. Patients with resectable disease but who refuse surgery may be enrolled after a documented consultation with a surgeon.
4. Radiologically or visually measurable disease that is at least 10mm in longest dimension, AND/OR with elevated disease specific serum markers that can be followed for progression (eg CA-125, AFP, PSA, CA19-9 or CEA)
5. ECOG performance status of ≤ 2.
6. Acceptable hematologic, renal and liver function as follows:

   A) Absolute neutrophil count > 1000/mm3 B) Platelets > 50,000/mm3, C) Creatinine ≤ 2.5 mg/dl, D) Total bilirubin ≤ 1.5 mg/dl, unless due to tumor or Gilbert's syndrome E) Transaminases ≤ 2 times above the upper limits of the institutional normal. F) INR<2 if off of anticoagulation. Patients on anticoagulation therapy with an INR>2 may be enrolled at the discretion of the investigator if they have not had any episodes of severe hemorrhage.
7. Patients must be able to provide informed consent.
8. Patients with the potential for pregnancy or impregnating their partner must agree to follow acceptable birth control methods to avoid conception. Contraception must be continued for at least 2 months following the last dose of Poly-ICLC. Women of childbearing potential must have a negative pregnancy test. While animal reproductive studies have been negative, the simulated viral infection and anti-proliferative activity of this experimental drug may theoretically affect the developing fetus or nursing infant.

   Cohort Specific Inclusion Criteria (see § 9.5 Evaluation of Best Overall Response (BOR)

   Cohort A
9. Patients who have received at least 8 weeks of immunotherapy.
10. Patients have progressive disease based on RECIST 1.1 criteria

    Cohort B)
11. Patients who have received at least 8 weeks of aPD1 or aPDL1 immunotherapy.
12. Patients have stable disease or a partial response based on RECIST 1.1 criteria.

    Cohort C)
13. Patients who have not received an anti-PD-1 or anti-PD-L1 agent, but who carry a diagnosis for which one of these agents is the SOC.
14. Patients willing to delay receipt of first dose of anti-PD-1 or anti-PD-L1 until after the receipt of their first two doses of intramuscular Poly-ICLC

Exclusion Criteria

1. Patients may not be receiving any other investigational agents.
2. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection requiring antibiotics (exception is a brief (≤10days) course of antibiotics to be completed before initiation of treatment), symptomatic congestive heart failure, unstable angina pectoris, or psychiatric illness/social situations that would limit compliance with study requirements.
3. Patients must not be pregnant or nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants.
4. Has a diagnosis of primary immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment. Patients on chronic steroids (more than 4 weeks at stable dose) equivalent to ≤ 10mg prednisone will not be excluded.
5. Has active autoimmune disease that has required systemic treatment in the past 1 year (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is acceptable.
6. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the patient's participation for the full duration of the trial, or is not in the best interest of the patient to participate, in the opinion of the treating Investigator.
7. HIV positive with detectable viral load, or anyone not on stable anti-viral (HAART) regimen, or with <200 CD4+ T cells/microliter in the peripheral blood.
8. Has known active Hepatitis B (e.g., HBV detected by elevated PCR or active Hepatitis C (e.g., HCV RNA [qualitative] is detected).
9. History of allogeneic hematopoietic cell transplantation or solid organ transplantation.
10. Documented allergic or hypersensitivity response to any protein therapeutics (e.g., recombinant proteins, vaccines, intravenous immune globulins, monoclonal antibodies, receptor traps)
11. Principal investigator believes that for one or multiple reasons the patient will be unable to comply with all study visits, or if they believe the trial is not clinically in the best interest of the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-09-25 (Actual); Primary Completion 2021-01-26 (Actual); Study Completion 2021-01-26 (Actual)

PRIMARY OUTCOMES:
Tumor assessment | 6 month timepoint compared to baseline
  Response and progression will be evaluated in this study. Tumor Response will be assessed by the RECIST 1.1 Criteria. Response is defined as CR, PR or SD over a period of at least 4 weeks. Changes in the sum of the two largest perpendicular diameters (SPD) of the tumor lesions, or the shortest diameter in the case of malignant lymph nodes are used in the RECIST 1.1 criteria. Study subjects with progressive disease will be evaluated to determine whether the progression causes symptoms and/or functional decline and study subjects with non-clinically relevant progression of disease may remain on study at the investigator's discretion.

CONTACTS AND LOCATIONS:
Overall Officials: Frederick P Smith, MD, Principal Investigator — Chevy Chase Healthcare; David H Smith, MD, Principal Investigator — Bay Hematology Oncology PA; Nina Bhardwaj, MD, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (3):
- United States (3):
  - Chevy Chase RCCA, Chevy Chase, Maryland
  - Bay Hematology Oncology, Easton, Maryland
  - Icahn School of Medicine at Mount Sinai, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bosio CM, Aman MJ, Grogan C, Hogan R, Ruthel G, Negley D, Mohamadzadeh M, Bavari S, Schmaljohn A. Ebola and Marburg viruses replicate in monocyte-derived dendritic cells without inducing the production of cytokines and full maturation. J Infect Dis. 2003 Dec 1;188(11):1630-8. doi: 10.1086/379199. Epub 2003 Nov 14. PMID 14639532
- [Result] Brody JD, Ai WZ, Czerwinski DK, Torchia JA, Levy M, Advani RH, Kim YH, Hoppe RT, Knox SJ, Shin LK, Wapnir I, Tibshirani RJ, Levy R. In situ vaccination with a TLR9 agonist induces systemic lymphoma regression: a phase I/II study. J Clin Oncol. 2010 Oct 1;28(28):4324-32. doi: 10.1200/JCO.2010.28.9793. Epub 2010 Aug 9. PMID 20697067
- [Result] Caskey M, Lefebvre F, Filali-Mouhim A, Cameron MJ, Goulet JP, Haddad EK, Breton G, Trumpfheller C, Pollak S, Shimeliovich I, Duque-Alarcon A, Pan L, Nelkenbaum A, Salazar AM, Schlesinger SJ, Steinman RM, Sekaly RP. Synthetic double-stranded RNA induces innate immune responses similar to a live viral vaccine in humans. J Exp Med. 2011 Nov 21;208(12):2357-66. doi: 10.1084/jem.20111171. Epub 2011 Nov 7. PMID 22065672